CLINICAL TRIAL: NCT03538847
Title: Postoperative Pain After Vitreo-retinal Surgery is Influenced by Duration of Surgery and Anaesthesia Conduction: a 1-year Retrospective Study.
Brief Title: Postoperative Pain After Vitreoretinal Surgery
Status: Completed | Type: Observational
Sponsor: University of Florence (Other)
Responsible Party: Principal Investigator, Dr. Chiara Adembri, Associate Professor, University of Florence
Other Study IDs: POP in VRS
Record Dates: First submitted 2018-05-04; First posted 2018-05-29 (Actual); Last update posted 2018-05-29 (Actual); Status verified 2018-05

CONDITIONS: Postoperative Pain; Retinal Detachment
Keywords: postoperative pain; eye surgery; vitrectomy; pain control protocol
MeSH Terms: conditions — Pain, Postoperative; Retinal Detachment

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Numerical rating scale — Measure of postoperative pain

SUMMARY:
Postoperative pain (POP) is frequently underestimated in general and little data are available particularly for POP after vitreoretinal surgery (VRS). The investigators will conduct a 1-year retrospective study on patients undergoing VRS at "Careggi Hospital" . The aim of the study will be to observe the amount of POP, its time course, factors associated with its appearance and finally the efficacy of the pain protocol that is in use.

DETAILED DESCRIPTION:
Post-operative pain (POP) is frequently underestimated, mostly after eye surgery, a type of surgery in which trauma is limited and pain is not investigated as patients are often discharged from the hospital within a few hours. Good POP management can improve clinical outcome and patients' satisfaction and constitutes essential criteria for hospital discharge after day-case or ambulatory surgery. Little data are available particularly for POP after vitreoretinal surgery (VRS).

The investigators will conduct a 1-year retrospective study on patients undergoing VRS at "Careggi Hospital" , a teaching University Hospital in Italy. The aim of the study will be to observe the amount of POP after VRS, its time course, factors associated with its appearance and finally the efficacy of the pain protocol that is in use.

Pain will be evaluated according to the "Numerical Rating Scale" (NRS), a 11-point numeric scale ranging from '0' which represents "no pain" and '10' which represents extreme pain at several intervals after surgery. Analgesic consumption (in terms of type and amount of analgesics) and the efficacy of the analgesic protocol in use will also be recorded.

Factors possibly associated with POP (such as duration of surgery, presence of comorbidities, ASA physical status, age, type of anesthesia (locoregional or general anesthesia)) will be analyzed.

The associations between the principal outcome (amount of POP) and risk factors will be evaluated using a simple and multiple logistic regression model.

ELIGIBILITY:
Inclusion Criteria:

* Vitreoretinal surgery

Exclusion Criteria:

* ASA IV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing vitreoretinal surgery under locoregional or general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2017-02-01 (Actual)

PRIMARY OUTCOMES:
postoperative pain | first day following surgery
  Numerical Rating Scale (NRS, a verbal numerical scale ranging from 0 to10, with 0 indicating no pain and 10 the maximal possible pain )

SECONDARY OUTCOMES:
age | day of surgery
  years
duration of surgery | day of surgery
  minutes
ASA (American Society of Anesthesiologists) PHYSICAL STATUS CLASSIFICATION SYSTEM I-IV (with I indicating a normal healthy patient and IV a patient with severe systemic disease that is a constant threat to life) | day of surgery
  I-IV (I : healthy patient; IV: worse state of health)
comorbidities | day of surgery
  presence
type of anesthesia | day of surgery
  general anesthesia
type of anesthesia | day of surgery
  locoregional anesthesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fekrat S, Marsh MJ, Elsing SH, Raja SC, de Juan E Jr, Campochiaro PA, Haller JA. Intraoperative ketorolac and eye pain after viteoretinal surgery: a prospective, randomized, placebo-controlled study. Retina. 2003 Feb;23(1):8-13. doi: 10.1097/00006982-200302000-00002. PMID 12652225
- [Background] Lesin M, Dzaja Lozo M, Duplancic-Sundov Z, Dzaja I, Davidovic N, Banozic A, Puljak L. Risk factors associated with postoperative pain after ophthalmic surgery: a prospective study. Ther Clin Risk Manag. 2016 Jan 22;12:93-102. doi: 10.2147/TCRM.S97024. eCollection 2016. PMID 26858525
- [Background] Ip HY, Abrishami A, Peng PW, Wong J, Chung F. Predictors of postoperative pain and analgesic consumption: a qualitative systematic review. Anesthesiology. 2009 Sep;111(3):657-77. doi: 10.1097/ALN.0b013e3181aae87a. PMID 19672167